CLINICAL TRIAL: NCT02825901
Title: Efficacy Testing of Djulis-Buckwheat Drink on Cardiovascular Protection
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to company policy, the development of this product is suspended.
Sponsor: Taipei Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: N201604003
Record Dates: First submitted 2016-06-14; First posted 2016-07-07 (Estimated); Last update posted 2023-11-22 (Actual); Status verified 2018-03

CONDITIONS: Prehypertension; Hypertension Stage 1
MeSH Terms: conditions — Prehypertension; Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Djulis-Buckwheat & Placebo (Active Comparator): Ingest Djulis-Buckwheat or placebo drink 100ml/day for 8 weeks
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: Djulis-Buckwheat
- Buckwheat & Placebo (Active Comparator): Ingest Buckwheat or placebo drink 100ml/day for 8 weeks
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: Buckwheat
- Djulis-Buckwheat & Buckwheat (Experimental): Ingest Djulis-Buckwheat or Buckwheat drink 100ml/day for 8 weeks
  Interventions: Dietary Supplement: Djulis-Buckwheat; Dietary Supplement: Buckwheat

INTERVENTIONS:
Dietary Supplement: Placebo — Ingest placebo drink 100ml/day for 8 weeks
  Arms: Buckwheat & Placebo; Djulis-Buckwheat & Placebo
Dietary Supplement: Djulis-Buckwheat — Ingest Djulis-Buckwheat drink 100ml/day for 8 weeks
  Arms: Djulis-Buckwheat & Buckwheat; Djulis-Buckwheat & Placebo
Dietary Supplement: Buckwheat — Ingest Buckwheat drink 100ml/day for 8 weeks
  Arms: Buckwheat & Placebo; Djulis-Buckwheat & Buckwheat

SUMMARY:
The purpose of the trial is to evaluate the effect of Djulis-Buckwheat drink on cardiovascular protection after ingesting for 8 weeks. In addition, the correlation between the supplement and the cardiovascular disease-related gene expression is evaluated. The results will be used for the application of functional products for cardiovascular protection.

Ninety subjects (age 30~65) with Prehypertension or Hypertension stage 1 will be included and randomly allocated into 3 groups: Placebo, Djulis-Buckwheat and Buckwheat. The subjects will take sample (100 ml/day) for 8 weeks. Blood pressure will be measured on week 0, 1, 2, 4, 6 and 8. The blood biochemical parameters and gene expression analysis will be examined on week 2, 4, 6, 8 and 10 (the follow up).

ELIGIBILITY:
Inclusion Criteria:

* Systolic blood pressure 121-159 mmHg or Diastolic blood pressure 81-99 mmHg
* Age: 30-65

Exclusion Criteria:

* Have diagnosed and documented critical illness(NHI specification)
* Had emergency record or admission note in the past three months
* Not be pregnant or breast-feeding a child

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Change of blood pressure | Baseline, 1, 2, 4, 6, and 8 weeks